CLINICAL TRIAL: NCT06397950
Title: Correlates of Fatigue in People With Schizophrenia
Acronym: FIZO-2
Status: Terminated | Type: Observational
Why Stopped: Recruitment difficulties caused by a lack of eligible patients in the investigating center, calling into question the feasibility of the study.
Sponsor: GCS CIPS (Other)
Responsible Party: Sponsor
Other Study IDs: FIZO-2
Record Dates: First submitted 2024-04-30; First posted 2024-05-03 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Schizophrenia
Keywords: Trait fatigue; Correlates; Physical activity; Sleep; Iatrogenic
MeSH Terms: conditions — Schizophrenia; Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with Schizophrenia: Patients are enrolled in a psychosocial rehabilitation program.
  Interventions: Other: Assessment of potential fatigue factors

INTERVENTIONS:
Other: Assessment of potential fatigue factors — 3 visits will be carried out: V0: Inclusion V1: Familiarization visit V2: Experimental visit
  V1
  * Completion of MFI-20 questionnaire for familiarisation.
  * Information about accelerometry and activity journal use will be delivered to the patient.
  * The participant will be equipped with an accelerometer and asked to complete the activity journal for seven days.
  V2
  * Completion of questionnaires: MFI-20, GATS tobacco consumption questionnaire, caffeine consumption questionnaire, Fatigue Catastrophizing Scale, PSQI.
  * Assessment of cognitive function: Sustained Attention to Response Task (SART), AX-Continuous Performance Task (AX-CPT) and verbal fluency test (animals and P categories).
  * Assessment of physical evaluation: isometric evaluation of maximal handgrip strength, one-minute sit-to-stand test, isometric evaluation of maximal quadriceps strength, QIF test.
  Negative symptoms will be assessed. Calf circumference will be measured for sarcopenia risk.

SUMMARY:
The goal of this experimental prospective study is to build an explicative model of trait fatigue in adults with schizophrenia engaged in a psychosocial rehabilitation process.

The main questions it aims to answer are:

* Which factors amongst those evaluated explain the most of fatigue variance in people with schizophrenia?
* Which clinical factors characterise the most fatigued participants compared to less fatigued participants?

Participants will wear an accelerometer for seven days to assess their sedentary and physical activity behaviours as well as their sleep.

After this, they will undergo an experimental visit, to asses:

* Fatigue
* Cognitive function
* Tobacco and caffeine consumption
* Fatigue catastrophizing
* Sleep quality
* Sarcopenia risk
* Functional capacities
* Handgrip strength
* Quadriceps maximal strength and fatigability

DETAILED DESCRIPTION:
Schizophrenia is a severe mental illness affecting about 1% of worldwide population. Diagnostic relies on multiple symptoms, divided into three main categories: positive symptoms, negative symptoms and cognitive/dissociative symptoms. Antipsychotic medication is actually the main pharmacologic treatment in schizophrenia but adverse effects can exacerbate other symptoms such as fatigue.

Fatigue has a high prevalence in schizophrenia. Unfortunately, fatigue has negative repercussions on daily living activities in this population, and no effective treatment has been identified for now. The lack of effective strategies to manage fatigue in schizophrenia can be due to the lack of knowledge about factors that can explain fatigue. As such, an explicative model of fatigue in schizophrenia has yet to be established.

Because fatigue is a complex and multifactorial mechanism, investigating its correlates could allow to propose new avenues for its multidisciplinary management, in order to delay its onset or minimize its negative impact. In comparison to healthy subjects, people with schizophrenia show increased physical inactivity and sedentary levels, worsened physical fitness and higher risks of sarcopenia, disturbed sleep, altered cognitive function, increased consumption of psychoactive substances (coffee and tobacco), an increased fatigue catastrophizing. Moreover, negative symptoms could also be linked to fatigue as it has been shown that fatigue could contribute to anhedonia in schizophrenia. Finally, antipsychotic medication can induce sedation, overlapping with fatigue, contributing to an exacerbated experience of the symptom.

Therefore, the goal of this study is to investigate whether physical inactivity, sedentary behaviour, physical fitness, sarcopenia risk, sleep, cognitive capacities, psychoactive substance consumption, fatigue catastrophizing, antipsychotic treatment and negative symptoms could contribute to fatigue in people in schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Patient with schizophrenia engaged in a psychosocial rehabilitation process.
* Patient with a stabilised evolution according to usual literature criteria (no modification or increase in antipsychotic treatment during the 4 weeks prior to inclusion).
* Absence of characterised major depressive episode.
* Patient affiliated or entitled to a social security scheme.
* Obtention of free and informed written consent, as well as the free and informed written consent of the guardian in the case of a patient placed under protection measure (guardianship).

Exclusion Criteria:

* Physical pain superior to 3 on a visual analog scale.
* History of severe inflammatory pathology or severe brain trauma.
* Medical contraindication to moderate-intensity physical activity practice.
* Patient having electroconvulsive therapy as current treatment.
* Addiction to toxic products such as alcohol, cannabis or other toxic substances other than tobacco.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be patients with schizophrenia, included in a psychosocial rehabilitation program.
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2024-10-11 (Actual); Primary Completion 2025-07-29 (Actual); Study Completion 2025-07-29 (Actual)

PRIMARY OUTCOMES:
Strength of predictive model of fatigue in schizophrenia | 8 days : 7 days for sleep, sedentary and physical activity levels recording, plus the experimental session (V2) for all other variables
  The aim is to determine the relative weight of the measured parameters to explain fatigue variance.
  * Fatigue score obtained at the MFI-20 will be selected as the dependent variable.
  * Muscle strength, muscle fatigue, functional abilities, risk of sarcopenia, sleep, cognition, antipsychotic treatment, smoking and coffee consumption, catastrophism, negative symptomatology, and physical activity and sedentary levels will be selected as independent variables.
  * Variables will be entered in a multiple linear regression to establish a predictive model of fatigue.

SECONDARY OUTCOMES:
Characterization of fatigued people with schizophrenia | 8 days : 7 days for sleep, sedentary and physical activity levels recording, plus the experimental session (V2) for all other variables
  The aim is to identify which clinical parameters characterize the most fatigued patients (F-group) compared to those who report less fatigue (NF-group)
  * Fatigued and less fatigued participants will be separated in two groups using the median score of the MFI-20 questionnaire as a cut point.
  * For each of the variables (muscle strength, muscle fatigue, functional abilities, risk of sarcopenia, sleep, cognition, antipsychotic treatment, smoking and coffee consumption, catastrophism, negative symptomatology, and physical activity and sedentary levels), comparison of means (Student T test or Mann-Whitney U test depending on application conditions) will be used to compare F-group to NF-group.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel MULIN, Principal Investigator — INICEA
Locations (1):
- Clinique INICEA Val Du Fenouillet, La Crau, France

IPD SHARING:
Plan to Share IPD: Undecided